CLINICAL TRIAL: NCT06662058
Title: Ototoxicity Monitoring and Remote Audiometry
Brief Title: Remote Audiometry to Monitor for Treatment-Related Hearing Loss in Patients With H&N SCC Receiving Cisplatin and/or Radiation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Nicole Schmitt, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008286; K24DC022077 (NIH); P30CA138292 (NIH); NCI-2024-08456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008286 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6359-24 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Head and Neck Carcinoma of Unknown Primary; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Metastatic Cutaneous Squamous Cell Carcinoma of the Head and Neck; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Nasopharyngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Metastatic Paranasal Sinus Squamous Cell Carcinoma; Nasopharyngeal Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Paranasal Sinus Squamous Cell Carcinoma; Recurrent Cutaneous Squamous Cell Carcinoma of the Head and Neck; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Nasopharyngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Paranasal Sinus Squamous Cell Carcinoma; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Sinonasal Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — Hearing; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (audiometry) (Active Comparator): Patients undergo audiometry at WEM at baseline and at 3 and 12 months after chemotherapy and/or radiation treatment.
  Interventions: Procedure: Audiometric Test; Other: Interview
- Group II, Arm I (audiometry) (Active Comparator): Patients undergo audiometry at WEM at baseline and at 3 and 12 months after chemotherapy and/or radiation treatment as in Group I.
  Interventions: Procedure: Audiometric Test; Other: Interview
- Group II, Arm II (close to home audiometry, remote audiometry) (Experimental): Patients undergo audiometry at WEM at baseline and are offered closer to home audiometry or self-administered remote audiometry at 3 and 12 months after chemotherapy and/or radiation treatment.
  Interventions: Procedure: Audiometric Test; Other: Interview

INTERVENTIONS:
Procedure: Audiometric Test — Undergo audiometry
  Other Names: Audiometric Testing; Audiometry; Hearing Test
Procedure: Audiometric Test — Undergo close to home audiometry
  Other Names: Audiometric Testing; Audiometry; Hearing Test
  Arms: Group II, Arm II (close to home audiometry, remote audiometry)
Procedure: Audiometric Test — Undergo self-administered remote audiometry
  Other Names: Audiometric Testing; Audiometry; Hearing Test
  Arms: Group II, Arm II (close to home audiometry, remote audiometry)
Other: Interview — Ancillary studies

SUMMARY:
This clinical trial tests the impact of offering hearing tests (audiometry) close to home and remotely on participation in monitoring for treatment-related hearing loss in patients with head and neck squamous cell cancer receiving cisplatin and/or radiation. Cisplatin, a chemotherapy often used to treat head and neck cancers, and radiation given near the ear can cause hearing loss in some patients. Hearing loss can have a major negative impact on quality of life, contributing to social isolation and frustration. Identifying hearing changes may allow treatment changes to prevent further loss. Audiometry measures hearing loss using a graphic record of the softest sounds that a person can hear at various frequencies. It is recommended patients have a hearing test before, during and after treatment to monitor for any hearing loss. This is usually done in the office and performed on the same day as other visits whenever possible, however, patients who live far away or have stage IV cancer, may have more difficulty coming back for hearing tests. Offering close to home and remote audiometry may improve monitoring for hearing loss in patients with head and neck squamous cell cancer receiving cisplatin and/or radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether a targeted intervention of remote audiometry offered to patients with advanced disease or living > 120 miles away increases overall participation in ototoxicity monitoring.

SECONDARY OBJECTIVE:

I. To estimate the incidence and severity of cisplatin-induced hearing loss in head and neck squamous cell carcinoma (HNSCC).

TERTIARY/EXPLORATORY OBJECTIVE:

I. To identify potential barriers to ototoxicity monitoring participation, from the patient perspective.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo audiometry at Winship Emory Midtown (WEM) at baseline and at 3 and 12 months after chemotherapy and/or radiation treatment.

GROUP II: Patients who do not live > 120 miles away or do not have stage IV disease are assigned to Arm I. Patients who do live > 120 miles away or who have stage IV disease are assigned to Arm II.

ARM I (USUAL): Patients undergo audiometry at WEM at baseline and at 3 and 12 months after chemotherapy and/or radiation treatment as in Group I.

ARM II (INTERVENTION): Patients undergo audiometry at WEM at baseline and are offered closer to home audiometry or self-administered remote audiometry at 3 and 12 months after chemotherapy and/or radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, aged ≥ 18, able to provide informed consent
* Subjects with pathologically proven HNSCC involving the oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, skin, or paranasal sinuses; patients with unknown primary HNSCC involving the cervical lymph nodes can also be included. Patients can have previously untreated or recurrent/metastatic disease
* Subjects who will be treated with cisplatin chemotherapy and/or radiation. For radiation alone, patients should have tumors near the inner ear, including the nasopharynx, temporal bone, and/or parotid salivary gland
* Life expectancy of more than 3 months, as determined by the investigator

Exclusion Criteria:

* Patients with profound hearing loss in both ears, which precludes an accurate hearing test. This can be determined based on patient report/history or audiogram done before or after informed consent
* Patients who are unable to participate in a hearing test (per the investigator's judgment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete at least one post-treatment audiogram | Up to 12 months post-treatment
  The incidence of follow-up audiometry relative to the targeted intervention will be assessed using a Z test for the equality of two proportions. An ordinal logistic regression analysis with mixed effects and calculations of odds ratios and 95% confidence intervals will be applied to identify associations between follow-up audiometry and intervention after adjustment for covariates including age, sex, race/ethnicity, pre-existing hearing loss, comorbidities, smoking, cisplatin dose (individual and cumulative) and cochlear radiation dose will be performed to assess whether the targeted intervention for at-risk patients is an independent predictor of increased overall participation.

SECONDARY OUTCOMES:
Incidence and severity of hearing loss | Up to 30 days following cessation of study participation
  Assessed using Common Terminology Criteria for Adverse Events criteria and American Speech Language and Hearing Association criteria.

OTHER OUTCOMES:
To identify potential barriers to ototoxicity monitoring participation | Up to 18 months post-treatment
  Qualitative data from patient interviews focused on barriers to ototoxicity monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole C Schmitt, MD, FACS, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory Midtown University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States